CLINICAL TRIAL: NCT02613208
Title: Observational and Prospective Study to Develop Predictive and Prognostic Tools for Optimizing Therapy With Bevacizumab Frontline Cancer Therapy in Patients With Metastatic HER 2-Negative and Aggressive Disease Criteria
Brief Title: A Study to Develop Predictive and Prognostic Tools for Optimizing Therapy With Bevacizumab Frontline Cancer Therapy in Participants With HER 2-Negative Aggressive Metastatic Breast Cancer
Acronym: Argo
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29756; ROC-BEV-2015-01 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Participants With Metastatic Breast Cancer: Participants with metastatic breast cancer receiving bevacizumab in combination with paclitaxel, will be observed for treatment responses for up to 18 months from the start of treatment.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered as per local clinical practice and local labeling.
Drug: Paclitaxel — Paclitaxel will be administered as per local clinical practice and local labeling.

SUMMARY:
This multicenter, observational, prospective study will identify a powerful and easy predictive/prognostic marker to use with participants under bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants with HER2-negative metastatic breast cancer. Mandatory to have the HER2/estrogen receptor (ER)/progesterone receptor (PR) status
* Participant who met criteria for first-line treatment with chemotherapy plus bevacizumab (standard doses) by local, regional or national guidelines or authorities
* Participants with measurable disease (RECIST criteria v1.1) or participants with no measurable but assessable disease
* Molecular phenotype as triple negative metastatic breast cancer; and ER-positive tumors need to fulfill at least one of the two clinical criteria: metastatic relapse on adjuvant endocrine therapy or progression to at least one prior line of endocrine therapy for advanced disease; or aggressive disease criteria (at least two criteria): taxane based regimen in the (neo) adjuvant setting; metastatic relapse within 2 years from the end of chemotherapy for early breast cancer; liver metastasis; three or more organs with metastatic involvement; symptomatic visceral disease
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Participant has received prior chemotherapy for metastatic disease
* Participant requiring major/minor surgery within 3 weeks prior to administration of the first dose of study treatment
* Participant has received an investigational therapy within 4 weeks prior to study entry
* Participant has known symptomatic brain metastases
* Participant with non-measurable or assessable disease: exclusive blastic bone disease; pleural, pericardial or abdominal effusion as only evidence of disease
* Participant in chronic daily treatment with corticosteroids (doses greater than [>]10 milligrams per day [mg/day] of methylprednisolone or equivalent), except inhaled steroids
* Pregnant or breastfeeding participant
* Women of childbearing potential who are not using hormonal contraceptives or highly effective birth control during the study
* Participant has an active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Participant with significant renal, hematological or liver function alteration according to investigator's criteria
* Participant has serious medical risk factors involving any of the major organ systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with human epidermal growth factor receptor 2 (HER2)-negative aggressive metastatic breast cancer treated with standard first line chemotherapy with paclitaxel-bevacizumab.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Spain (25):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital de Donostia.; Servicio de Oncología Radioterápica, San Sebastián, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Oncologia, A Coruña, LA Coruña
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Quiron Barcelona; Servicio de Oncologia, Barcelona
  - Hospital Universitario Virgen de las Nieves; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - Hospital Universitario de la Princesa; Servicio de Oncologia, Madrid
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital General de Segovia; Servicio de Oncologia, Segovia
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Oncologia, Valencia
  - Complejo Hospitalario Zamora- H. Virgen de la Concha; Servicio Oncologia, Zamora

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Metastatic Breast Cancer
Started | 111
Completed | 64
Not Completed | 47
Not completed — Withdrawal by Subject | 1
Not completed — Change of address | 2
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 5
Not completed — Death | 37

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Race : Caucasian | 105
  Race : Latino | 4
  Race : Black | 1
  Race : Arab | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). Clinical benefit is defined as partial or complete response as well as tumor stabilization for up to 24 weeks. Results for clinical benefit were reported for 2 groups based on Circulating Tumor Cells (CTC) Levels. The Sensitive group had CTC levels <5 (<5 CTCs in one of the two determinations) and Resistant group had CTC ≥5 (≥ 5 CTCs in the two determinations).
Time Frame: During follow-up (up to 18 months)
Population: Included participants that were evaluable for CTC level after cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
Participants
  Sensitive: number analyzed (Participants) | 73
  Sensitive: Benefit = Yes | 53
  Sensitive: Benefit = No | 20
  Resistant: number analyzed (Participants) | 12
  Resistant: Benefit = Yes | 5
  Resistant: Benefit = No | 7

2. Secondary Outcome: Percentage of Participants With Overall Response as Assessed Using RECIST v1.1
Description: Overall response = Complete Response (CR) + Partial Response (PR). Overall response was evaluated for the Sensitive group (CTC <5) and Resistant group (CTC ≥5).
Time Frame: From Baseline up to end of study (up to 18 months)
Population: Included participants that were evaluable for CTC level after cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
Participants
  Sensitive: number analyzed (Participants) | 73
  Sensitive: Overall Response = Yes | 35
  Sensitive: Overall Response = No | 38
  Resistant: number analyzed (Participants) | 12
  Resistant: Overall Response = Yes | 2
  Resistant: Overall Response = No | 10

3. Secondary Outcome: Progression Free Survival (PFS) as Assessed Using RECIST v1.1
Description: PFS was evaluated for the Sensitive group (CTC <5) and Resistant group (CTC ≥5).
Time Frame: From Baseline up to end of study (up to 18 months)
Population: Included participants that were evaluable for CTC level after cycle 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
months
  Sensitive: number analyzed (Participants) | 73
  Sensitive | 17.38 [15.15 to 19.06]
  Resistant: number analyzed (Participants) | 12
  Resistant | 5.49 [2.97 to 8.00]

4. Secondary Outcome: Overall Survival
Description: OS was evaluated for the Sensitive group (CTC <5) and Resistant group (CTC ≥5).
Time Frame: From Baseline up to end of study (up to 18 months)
Population: Included only participants that were evaluable for CTC level after cycle 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
months
  Sensitive: number analyzed (Participants) | 73
  Sensitive | NA [NA to NA] — Median OS in patients with CTCs <5 was not achieved
  Resistant: number analyzed (Participants) | 12
  Resistant | 13.01 [5.82 to 20.20]

5. Secondary Outcome: Percentage of Participants With Adverse Events of Toxicity Grading 3 and/or 4
Description: Adverse events (AEs) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v 4.0). Any AEs that are not specifically listed in the NCI CTCAE follow the logic - Grade 3) Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4: Life-threatening consequences or urgent intervention indicated.
Time Frame: From Baseline up to end of study (up to 18 months)
Population: Included only participants that were evaluable for CTC level after cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
Participants
  Sensitive: number analyzed (Participants) | 73
  Sensitive: Grade 3-4 toxicity = yes | 28
  Sensitive: Grade 3-4 toxicity = no | 45
  Resistant: number analyzed (Participants) | 12
  Resistant: Grade 3-4 toxicity = yes | 6
  Resistant: Grade 3-4 toxicity = no | 6

6. Secondary Outcome: Optimal Cut-off for Clinical Benefit
Description: Clinical benefit was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). Clinical benefit is defined as partial or complete response as well as tumor stabilization for up to 24 weeks. The optimal cut-off for clinical benefit was calculated from a Receiver Operating Curve (ROC) based on CTC level and used to define the prognostic factors that could better predict clinical outcomes.
Time Frame: Baseline (within 21 days prior to Day 1 Cycle 1), 7 days prior to Day 1 Cycle 3 (Cycle length = 28 days)
Population: Included only participants that were evaluable for CTC level after cycle 2.
Measure: Number; unit: cells/7.5 ml
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
cells/7.5 ml | 0.5

7. Secondary Outcome: Percentage of Participants With Overall Response (OR) as Assessed Using RECIST v1. in Prognostic Groups
Description: Overall response = CR + PR. An optimal cut-off point for the CTC count of 0.5 after 2 cycles of treatment was used to define the prognostic groups.
Time Frame: Baseline (within 21 days prior to Day 1 Cycle 1), 7 days prior to Day 1 Cycle 3 (Cycle length = 28 days)
Population: Included only participants that were evaluable for CTC level after cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
Participants
  CTC >0.5: number analyzed (Participants) | 41
  CTC >0.5: Overall Response = Yes | 14
  CTC >0.5: Overall Response = No | 27
  CTC ≤0.5: number analyzed (Participants) | 44
  CTC ≤0.5: Overall Response = Yes | 23
  CTC ≤0.5: Overall Response = No | 21

8. Secondary Outcome: PFS as Assessed Using RECIST v1. in Prognostic Groups
Description: An optimal cut-off point for the CTC count of 0.5 after 2 cycles of treatment was used to define the prognostic groups.
Time Frame: From Baseline up to end of study (up to 18 months)
Population: Included only participants that were evaluable for CTC level after cycle 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 85
months
  CTC <0.5: number analyzed (Participants) | 44
  CTC <0.5 | 22.60 [NA to NA] — Not estimable due to insufficient number of participants with events.
  CTC ≥0.5: number analyzed (Participants) | 41
  CTC ≥0.5 | 8.05 [5.35 to 10.75]

9. Secondary Outcome: Mean CTC Count Levels
Description: CTC and CEA levels were compared to determine any correlation between the two. Both CTC count at baseline and at cycle 2 were considered.
Time Frame: Baseline (within 21 days prior to Day 1 Cycle 1 [Cycle length = 28 days])
Population: Only included participants that had available data of CTC levels at baseline
Measure: Mean (Standard Deviation); unit: count/7.5 ml (CTC)
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 89
count/7.5 ml (CTC)
  CTC (baseline CTC): number analyzed (Participants) | 87
  CTC (baseline CTC) | 91.6 (355.5)
  CTC (cycle 2 CTC): number analyzed (Participants) | 85
  CTC (cycle 2 CTC) | 3.9 (10.8)
Statistical Analysis 1: Comparison: Participants With Metastatic Breast Cancer; Correlation between CTC and CEA level considering baseline CTC count; Test type: Other — Correlation analysis; p < 0.001, Spearman's correlation analysis; Spearman coefficient = 0.392
Statistical Analysis 2: Comparison: Participants With Metastatic Breast Cancer; Correlation between CTC and CEA level considering CTC count at cycle 2; Test type: Other — Correlation analysis; p = 0.444, Spearman's correlation analysis; Spearman coefficient = 0.088

10. Secondary Outcome: Mean Carcinoembryonic Antigen (CEA) Levels
Time Frame: Baseline (within 21 days prior to Day 1 Cycle 1 [Cycle length = 28 days])
Population: Only included participants that had available data of CEA levels at baseline
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 89
U/ml | 46.5 (146.2)

11. Secondary Outcome: Mean Biomarker Cancer Antigen 15.3 (CA 15.3) Level
Description: CTC and CA 15.3 levels were compared to determine any correlation between the two. Both CTC count at baseline and at cycle 2 were considered.
Time Frame: Baseline (within 21 days prior to Day 1 Cycle 1 [Cycle length = 28 days])
Population: Only included participants that had available data of CA 15.3 levels at baseline
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 95
U/ml | 277.8 (431.3)
Statistical Analysis 1: Comparison: Participants With Metastatic Breast Cancer; Correlation between CTC and CA 15.3 level considering baseline CTC count; Test type: Other — Correlation analysis; p < 0.001, Spearman's correlation analysis; Spearman coefficient = 0.373
Statistical Analysis 2: Comparison: Participants With Metastatic Breast Cancer; Correlation between CTC and CA 15.3 level considering CTC count at cycle 2; Test type: Other — Correlation analysis; p = 0.241, Spearman's correlation analysis; Spearman coefficient = 0.129

ADVERSE EVENTS:
Time Frame: From Baseline up to end of study (up to 18 months)
Arm/Group | Participants With Metastatic Breast Cancer
All-Cause Mortality (participants affected / at risk) | 37/111
Serious Adverse Events (participants affected / at risk) | 37/111
Other Adverse Events (participants affected / at risk) | 107/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Metastatic Breast Cancer (N=111)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
DIPLOPIA (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
ENTERITIS (Gastrointestinal disorders) | 1
GASTRIC PERFORATION (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
DISEASE PROGRESSION (General disorders) | 1
FATIGUE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2
MUCOSAL INFLAMMATION (General disorders) | 1
PYREXIA (General disorders) | 1
VASCULAR DEVICE INFECTION (General disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
ABDOMINAL SEPSIS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
UROSEPSIS (Infections and infestations) | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
CONFUSIONAL STATE (Nervous system disorders) | 1
EXTRAOCULAR MUSCLE PARESIS (Nervous system disorders) | 1
URINARY TRACT INFECTION (Renal and urinary disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1
PULMONARY EMBOLISM (Vascular disorders) | 1
SUBDURAL HAEMATOMA (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Metastatic Breast Cancer (N=111)
ANAEMIA (Blood and lymphatic system disorders) | 23
NEUTROPENIA (Blood and lymphatic system disorders) | 18
ABDOMINAL PAIN (Gastrointestinal disorders) | 9
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6
CONSTIPATION (Gastrointestinal disorders) | 23
DIARRHOEA (Gastrointestinal disorders) | 41
DYSGEUSIA (Gastrointestinal disorders) | 6
GINGIVAL BLEEDING (Gastrointestinal disorders) | 9
NAUSEA (Gastrointestinal disorders) | 29
STOMATITIS (Gastrointestinal disorders) | 11
TOOTHACHE (Gastrointestinal disorders) | 7
VOMITING (Gastrointestinal disorders) | 17
ASTHENIA (General disorders) | 51
CHEST PAIN (General disorders) | 7
FATIGUE (General disorders) | 25
INFUSION RELATED REACTION (General disorders) | 7
MUCOSAL INFLAMMATION (General disorders) | 12
PAIN (General disorders) | 6
PYREXIA (General disorders) | 18
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 9
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 6
NEUTROPHIL COUNT DECREASED (Investigations) | 15
PLATELET COUNT DECREASED (Investigations) | 11
DECREASED APPETITE (Metabolism and nutrition disorders) | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 12
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14
DIZZINESS (Nervous system disorders) | 7
HEADACHE (Nervous system disorders) | 18
NEUROPATHY PERIPHERAL (Nervous system disorders) | 22
NEUROTOXICITY (Nervous system disorders) | 18
PARAESTHESIA (Nervous system disorders) | 15
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8
POLYNEUROPATHY (Nervous system disorders) | 15
ANXIETY (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 6
PROTEINURIA (Renal and urinary disorders) | 9
URINARY TRACT INFECTION (Renal and urinary disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 14
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 13
UPPER RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 6
ALOPECIA (Skin and subcutaneous tissue disorders) | 35
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 8
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 15
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 12
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 25
RASH (Skin and subcutaneous tissue disorders) | 12
EPISTAXIS (Vascular disorders) | 48
HYPERTENSION (Vascular disorders) | 48
RECTAL HAEMORRHAGE (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02613208/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT02613208/SAP_001.pdf